CLINICAL TRIAL: NCT07259876
Title: Efficacy and Neurophysiological Correlates of a Bilateral Robotic Treatment for the Upper Limbs in Patients With Chronic Stroke Outcomes
Brief Title: Efficacy of a Bilateral Robotic Treatment in Chronic Patients
Acronym: BUILT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); Centro Riabilitativo Villa Beretta (Unknown); Fondazione Don Carlo Gnocchi Onlus (Other); Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Carmelo Chisari, Professor, University of Pisa
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0017901/2025
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left hemisphere lesion group (Experimental): The stroke patients with left hemisphere lesion will be performing the bilateral robotic treatment with the exoskeleton ALEx-RS followed by a standard manual treatment
  Interventions: Device: Bilateral robotic treatment for the upper limbs; Behavioral: Standard physiotherapy
- Right hemisphere lesion group (Experimental): The stroke patients with right hemisphere lesion will be performing the bilateral robotic treatment with the exoskeleton ALEx-RS followed by a standard manual treatment
  Interventions: Device: Bilateral robotic treatment for the upper limbs; Behavioral: Standard physiotherapy

INTERVENTIONS:
Device: Bilateral robotic treatment for the upper limbs — Patients will perform a specific sequence of exercises with the exoskeleton for the upper limbs ALEx-RS, including passive and active-assisted movements, unilateral and bilateral reaching tasks with visual feedback, and symmetric and asymmetric bimanual coordination tasks.
Behavioral: Standard physiotherapy — After the robotic treatment, patients will undergo 20 minutes of conventional treatment consisting of passive and active-assisted mobilization with the help of a physiotherapist.

SUMMARY:
The goal of this clinical trial is to evaluate how manual dominance influences the effectiveness of bilateral robotic treatment in right-handed patients with chronic stroke.

Researchers will compare the outcome of a bilateral robotic treatment for the upper limbs in left vs right hemisphere lesions following stroke.

Participants will:

* perform a bilateral robotic treatment for the upper limb (15 sessions in three weeks) followed by 20-minutes standard manual rehabilitative sessions
* be evaluated before and after treatment with clinical scales, resting- state EEG and kinematic measurements

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 80 years, of either sex
* Subjects able to understand and provide, or have provided on their behalf, informed consent
* History of a single unilateral ischemic or hemorrhagic cerebrovascular event in the chronic phase (> 6 months)
* Subjects with mild to moderate functional impairment of the right or left upper limb (ability to perform antigravity active movements)

Exclusion Criteria:

* Subjects with cognitive deficits that impair understanding of the required tasks (MMSE score corrected for age and education < 24/30)
* Subjects with severe visual deficits
* Subjects with upper limb spasticity preventing the use of robotic devices (spasticity measured using the Modified Ashworth Scale > 3)
* Inability or unwillingness to provide informed consent
* Left-handed subjects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Fugl-Meyer for the upper limb functional scale (UEFM) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 66, with higher scores indicating better performance

SECONDARY OUTCOMES:
Changes in the Bimanual Activity Test scale (BAT) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 100, with higher scores indicating better performance
Changes in the modified Ashworth scale (MAS) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 6, with lower scores indicating better performance
Changes in the Stroke Impact Scale (SIS) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 100, with higher scores indicating better performance
Changes in the Visual Analogue Scale (VAS) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 10, with higher scores indicating higher pain
Changes in the Quick Dash scale | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The scale ranges from 0 to 100, with higher scores indicating higher level of disability
Changes in weighted Phase Lag Index (wPLI) cortico-cortical brain connectivity (EEG) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The investigators will be measuring variations in the weighted Phase Lag Index (wPLI)
Changes in weighted Symbolic Mutual Information (wSMI) cortico-cortical brain connectivity (EEG) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The investigators will be measuring variations in the weighted Symbolic Mutual Information (wSMI)
Changes in muscular synergies (EMG) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The investigators wil be measuring changes in muscle synergy patterns using the non-negative matrix factorization (NMF) algorithm
Changes in kinematic movement smoothness (SPARC) | From the pre-training evaluation (T0) to the follow up (T2), about 11 weeks after T0
  The investigators will measure changes in movement smoothness using the SPARC parameter

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication